CLINICAL TRIAL: NCT04024982
Title: The Ideal Sequence of Didactic Lectures and Simulation in Teaching Transoesophageal Echocardiography (TEE) Among Anaesthesiologists
Brief Title: TEE Training for Anaesthesiologists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, NUS Anaesthesia, Principal Investigator, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NUS IRB S-17-347
Record Dates: First submitted 2019-07-15; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Cardiac
Keywords: Transoesophageal Echocardiography (TEE); Learning

STUDY DESIGN:
Intervention Model Description: The TEE session will consist of a 1-hour lecture and a 2-hour simulation session. Participants for the TEE session are divided into 2 groups. Trainee participants are randomly divided into groups A and B. The specialists are also randomly divided into groups C and D. Groups A and C undergo lecture first then simulation, whereas B and D undergo simulation first then lecture.
  Prior to the teaching session (lecture or simulation), the participants will take a MCQ pre-test with 30 questions relating to TEE safety, probe manipulation and basic views in TEE. There is no pre-test on technical skill, as all of them are novices to TEE (i.e. with no skill on TEE). A post-test consisting of 30 MCQs (same as pre-test but in a different sequence) and a technical skill test is held at the completion of both lecture and simulation sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lecture followed by Simulation (Other): Subjects will undergo the lecture on TEE first followed by the simulation session.
  Interventions: Other: Sequence of teaching (Lecture first followed by Simulation)
- Simulation followed by Lecture (Other): Subjects will undergo the TEE simulation first followed by the lecture.
  Interventions: Other: Sequence of teaching (Simulation first followed by Lecture)

INTERVENTIONS:
Other: Sequence of teaching (Lecture first followed by Simulation) — Sequence of teaching (whether lecture or simulation session first) can help to achieve the maximum skill acquisition in TEE.
  Arms: Lecture followed by Simulation
Other: Sequence of teaching (Simulation first followed by Lecture) — Sequence of teaching (whether lecture or simulation session first) can help to achieve the maximum skill acquisition in TEE.
  Arms: Simulation followed by Lecture

SUMMARY:
This study aims to find out the best sequence of teaching and learning events (i.e. first lecture and then simulated training or first simulated training and then lecture) in the acquisition of knowledge on Transoesophageal Echocardiography among trainee and specialist anaesthesiologists.

DETAILED DESCRIPTION:
Basic Transoesophageal Echocardiography (TEE) is an essential skill in the armamentarium of an anaesthesiologist. Currently, majority of the TEE teaching is being done in the form of didactic lectures with only a few teaching centres offering simulation. TEE skill acquisition includes both technical and cognitive skills. Most of the studies done in TEE teaching have concluded that TEE simulation is an essential part of TEE skill training. The study team wanted to find out what is the best sequence of teaching to achieve the maximum skill acquisition in TEE.

In National University Hospital, Singapore, the Cardiac subdivision of anaesthesia specialists are accredited in TEE (American or European exams) and perform independent decision making in cardiac surgical theatres while the surgery is on-goingto facilitate dynamic decision making such as adequacy of valve repair, global LV function and emerging complications if any. The study team realised that TEE skills are also required for decisions beyond the cardiac surgical theaters where on the spot critical decisions making is required eg: in polytrauma and sudden unexplained hypotension or hypoxia in non-cardiac or ICU patients.

There are existing induction modules and prior teaching avenues in the department of anaesthesia such as the Cardiac Anaesthesia Simulation Training (CAST) module targeted at junior trainee's level. With initiative to equip every practicing anaesthesiologist with the vital skill of TEE image acquisition, the department of anaesthesia is launching a teaching program that is an in house training session. The study team aims to understand through this study the ideal sequence of teaching intervention to facilitate optimal learning and retention.

ELIGIBILITY:
Inclusion Criteria:

* All anaesthesia doctors in Singapore with no prior experience in TEE.

Exclusion Criteria:

* All anaesthesia doctors in Singapore with prior experience in TEE.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-11-17 (Actual); Study Completion 2018-11-17 (Actual)

PRIMARY OUTCOMES:
Knowledge and skill increment between both groups | Within an hour of completion of both lecture and simulation sessions.
  After the end of both lecture and simulation session, participants will be asked to demonstrate skill of acquisition of 11 basic views on TEE simulator within stipulated time, and will be scored by 2 independent raters.

SECONDARY OUTCOMES:
Demographic variations in knowledge and skill acquisition | Within an hour of completion of both lecture and simulation sessions.
  Identify and compare whether there are demographic variations in knowledge and skill acquisition in TEE among anaesthesiologists within each sequence of teaching and learning (i.e. lecture followed by simulation training and simulation training followed by lecture). This will be done through the administration of 30-question MCQ relating to TEE safety, probe manipulation and basic views in TEE, and a technical skill test.

CONTACTS AND LOCATIONS:
Overall Officials: Swapna Thampi, Principal Investigator — National University Health System
Locations (1):
- National University Health System, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No